CLINICAL TRIAL: NCT05306184
Title: Prospective Assessment of Cost-effectiveness and Side-effects of Depressive Patients Treated With ECT or TCA
Acronym: PROSPECT
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: GGZ inGeest (Other); Canisius-Wilhelmina Hospital (Other); UMC Utrecht (Other); St. Antonius Hospital (Other); ETZ (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-13224
Record Dates: First submitted 2022-03-20; First posted 2022-04-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive disorder; ECT; Electroconvulsive therapy; Antidepressants; Cost-effectiveness
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECT group: 110 participants with primary diagnosis of moderate to severe major depressive disorder receiving ECT as treatment
  Interventions: Procedure: Electroconvulsive therapy (ECT)
- Medication group: 110 participants with primary diagnosis of moderate to severe major depressive disorder receiving medication as treatment

INTERVENTIONS:
Procedure: Electroconvulsive therapy (ECT) — ECT
  Groups: ECT group

SUMMARY:
Prospective observational cohort study to determine cost-effectiveness of ECT compared to medication in the treatment of major depressive disorder (MDD) in the Netherlands.

DETAILED DESCRIPTION:
Rationale:

Currently, detailed information on the cost-effectiveness of ECT based on real-world data is lacking, as well as the comparative cost-effectiveness with respect to medication. Reliable information on outcomes of ECT in comparison with antidepressant treatment and its cognitive side-effects is needed for patients and clinicians to make a balanced and shared decision regarding choosing or refraining from ECT.

Objective:

Primary Objective: determine (cost)-effectiveness of ECT compared to medication by determining the impact of treatment for MDD with ECT or TCA on remission rates using a one-year time horizon (trial-based economic evaluation)

Secondary Objective: determine side-effects of ECT compared to medication by determining the impact of treatment with ECT or medication on side-effects and quality of life during a one-year follow-up

Study design: Observational, parallel inception cohort study of patients who will undergo standard clinical care according to current guidelines.

Study population: 110 patients (>18 yrs.) with a depressive episode (unipolar MDD) who will start ECT (ECT group) and 110 patients (>18 yrs.) with a depressive episode (unipolar MDD) who will undergo treatment with antidepressants will be recruited from specialized clinics (academic hospital, general hospital and GGz-institute) and followed-up for one year to gather reliable data on efficacy including relapse rates, cost-effectiveness, quality of life and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years) with a major depressive disorder who will either start with ECT or medication
* failed response to at least 1 adequate dose-duration trial with antidepressants
* moderate or severe depression (HDRS-17 >16)

Exclusion Criteria:

* lifetime diagnosis schizophrenia or schizoaffective disorder, current substance abuse disorder, organic brain syndrome
* the presence of a concurrent significant medical condition impeding the ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 110 patients (>18 yrs.) with a depressive episode (unipolar MDD) who will start ECT and 110 patients (>18 yrs.) with a depressive episode (unipolar MDD) who will undergo treatment with antidepressants will be recruited from specialized clinics (academic hospital, general hospital and GGz-institute) and followed-up for one year to gather reliable data on efficacy including relapse rates, cost-effectiveness and quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of treatment as measured by reduction on HDRS-17 | change from baseline at 3 months, 6 months and 12 months
  Depression severity measured by The Hamilton Depression Rating Scale 17 item version (HDRS-17)

SECONDARY OUTCOMES:
Cost-effectiveness as measured with The Trimbos Institute and iMTA Cost questionnaire for Psychiatry (TiC-P) | change from baseline at 3 months, 6 months and 12 months
  Cost-effectiveness as measured with The Trimbos Institute and iMTA Cost questionnaire for Psychiatry (TiC-P)
Quality of life as measured with the EuroQol-5D (EQ-5D-5L) | change from baseline at 3 months, 6 months and 12 months
  Quality of life as measured with the EuroQol-5D (EQ-5D-5L)
Cognitive functioning as measured by Montreal Cognitive Assesment (MoCA) | change from baseline at 3 months, 6 months and 12 months
  Cognitive functioning as measured by Montreal Cognitive Assesment (MoCA)
COLUMBIA UNIVERSITY - AUTOBIOGRAPHICAL MEMORY INTERVIEW SHORT FORM (CU-AMI-SF) | change from baseline at 3 months, 6 months and 12 months
Subjective Assessment of Memory Impairment (SAMI) | change from baseline at 3 months, 6 months and 12 months
  Subjective Assessment of Memory Impairment (SAMI)
15 words test (15WT) | change from baseline at 3 months, 6 months and 12 months
  (15WT; Saan & Deelman, 1986)
Verbal fluency test (e.g., Lezak et al., 2012). | change from baseline at 3 months, 6 months and 12 months
  It typically consists of two tasks: category fluency (sometimes called semantic fluency; Benton, 1968) and letter fluency (sometimes called phonemic fluency; Newcombe, 1969). participants are given 1 min to produce as many unique words as possible within a semantic category (category fluency) or starting with a given letter (letter fluency).

CONTACTS AND LOCATIONS:
Overall Officials: Philip van Eijndhoven, PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - GGz inGeest, Amsterdam
  - RadboudUMC, Nijmegen

IPD SHARING:
Plan to Share IPD: No